CLINICAL TRIAL: NCT00341874
Title: Genetic Analyses of Nonsyndromic and Syndromic Deafness in Pakistan
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999993016; OH93-DC-016
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-10-06

CONDITIONS: Hearing Disorder
Keywords: DNA Mutations; Genetic Variations; GENETIC LINKAGE; Usher Syndrome; BLINDNESS; Natural History
MeSH Terms: conditions — Hearing Disorders; Usher Syndromes; Blindness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Subjects with hearing loss consisting of both nonsyndromic and syndromic forms of deafness of genetic etiology

SUMMARY:
Objective: One objective of this study is to genetically map and identify mutated genes for human hereditary hearing loss. A second objective is to study the function of these genes in the auditory system using mouse models. Human hereditary hearing impairment is the result of abnormal ear development, abnormal ear function or both. Although the genes for numerous deafness loci have been mapped and identified, there are still many families segregating deafness as a monogenic trait but a mutant allele can t be ascribed to one of the currently reported deafness genes . In order to map and identify novel mutated genes associated with hearing loss in humans, we will continue to ascertain large families segregating syndromic and nonsyndromic deafness as a monogenic trait.

Study population: This study will ascertain subjects from consanguineous Pakistani families segregating hearing loss consisting of both nonsyndromic and syndromic forms of deafness of genetic etiology. Since a majority of Pakistani marriages are between first cousins, this tends to bring together the same recessive mutations for hearing loss with multiple affected individuals within single family lines, which is an advantage for this genetic study. A few years ago we stopped ascertaining families in India. We continue to ascertain both affected and unaffected Pakistani family members from age 2 years and up. Adults provide informed consent both for themselves and their children who agree to participate in this study. We will ascertain both genders and all Pakistani races and ethnicities.

Design: Subjects will be screened and consented by our collaborating Associate Investigator in Pakistan. After consenting, the subjects will undergo a history and physical, audiological assessment and testing, vestibular assessment and testing, and blood and urine analysis tests, along with a blood sample or buccal swab sample that will be used for genomic DNA extraction. Probands at the time of ascertainment are initially assumed to have a form of nonsyndromic deafness. Additional tests may be performed depending on the history or physical of the individual or after the deafness gene is identified. Data from functional studies in animal models may also point to other concomitant clinical features along with hearing loss. These additional tests may include: photographs or videotapes of a subject s body and face; eye and vision examinations for those with suspected or known eyesight problems related to their genetic hearing loss mutations, and EKGs and/or Echocardiograms for those with suspected or known heart problems related to their genetic hearing loss mutations. Urine and blood analyses may be requested for those individuals with genetic nephritic issues or infertility. For example, when a deaf female individual in a family is subsequently discovered to have Perrault syndrome, a recessive disorder characterized by hearing loss (usually the initial manifestation) and ovarian dysgenesis/primary amenorrhea, additional evaluations would then be conducted for a definitive diagnosis of Perrault syndrome. Such an evaluation would include a pelvic ultrasound scan and measurements of serum estrogen and gonadotropins. Similarly, in some of these families, hearing impaired males may be asked about their fertility since the possibility of male infertility in families segregating Perrault syndrome remains an open question. For genetic analyses, genomic DNA extracted from a blood sample or a buccal swab from affected and unaffected members of families segregating hereditary hearing loss will be genetically screened with polymorphic markers (STRs or SNPs) for linkage to the known deafness loci. The hearing phenotype of children (>2 years old), adolescent and adult subjects will be assigned on the basis of performance from audiological examinations. Genomic DNA from families where deafness is found to be unlinked to the known deafness loci will then be used in genome wide screens with approximately 950,000 SNP markers distributed across the entire human genome to identify novel deafness loci. Alternatively, DNA samples from affected and unaffected individuals will undergo whole exome sequencing (WES) or whole genome sequencing (WGS) with a focus on potentially pathogenic variants located only in chromosomal regions of markers genetically linked to deafness. Subsequently, novel deafness genes will be positionally identified and their functions studied.

Outcome measures: Novel deafness loci and genes associated with hearing loss will be identified and will provide new insight into mechanisms required for sound transduction in humans. Data from this study is likely to be the basis of commercially available tests for early diagnosis and timely genetic counseling for at risk couples as well as the development of strategies to preserve hearing and prevent hearing loss.

DETAILED DESCRIPTION:
Objective: One objective of this study is to genetically map and identify mutated genes for human hereditary hearing loss. A second objective is to study the function of these genes in the auditory system using mouse models. Human hereditary hearing impairment is the result of abnormal ear development, abnormal ear function or both. Although the genes for numerous deafness loci have been mapped and identified, there are still many families segregating deafness as a monogenic trait but a mutant allele can t be ascribed to one of the currently reported deafness genes . In order to map and identify novel mutated genes associated with hearing loss in humans, we will continue to ascertain large families segregating syndromic and nonsyndromic deafness as a monogenic trait.

Study population: This study will ascertain subjects from consanguineous Pakistani families segregating hearing loss consisting of both nonsyndromic and syndromic forms of deafness of genetic etiology. Since a majority of Pakistani marriages are between first cousins, this tends to bring together the same recessive mutations for hearing loss with multiple affected individuals within single family lines, which is an advantage for this genetic study. A few years ago we stopped ascertaining families in India. We continue to ascertain both affected and unaffected Pakistani family members from age 2 years and up. Adults provide informed consent both for themselves and their children who agree to participate in this study. We will ascertain both genders and all Pakistani races and ethnicities.

Design: Subjects will be screened and consented by our collaborating Associate Investigator in Pakistan. After consenting, the subjects will undergo a history and physical, audiological assessment and testing, vestibular assessment and testing, and blood and urine analysis tests, along with a blood sample or buccal swab sample that will be used for genomic DNA extraction. Probands at the time of ascertainment are initially assumed to have a form of nonsyndromic deafness. Additional tests may be performed depending on the history or physical of the individual or after the deafness gene is identified. Data from functional studies in animal models may also point to other concomitant clinical features along with hearing loss. These additional tests may include: photographs or videotapes of a subject s body and face; eye and vision examinations for those with suspected or known eyesight problems related to their genetic hearing loss mutations, and EKGs and/or Echocardiograms for those with suspected or known heart problems related to their genetic hearing loss mutations. Urine and blood analyses may be requested for those individuals with genetic nephritic issues or infertility. For example, when a deaf female individual in a family is subsequently discovered to have Perrault syndrome, a recessive disorder characterized by hearing loss (usually the initial manifestation) and ovarian dysgenesis/primary amenorrhea, additional evaluations would then be conducted for a definitive diagnosis of Perrault syndrome. Such an evaluation would include a pelvic ultrasound scan and measurements of serum estrogen and gonadotropins. Similarly, in some of these families, hearing impaired males may be asked about their fertility since the possibility of male infertility in families segregating Perrault syndrome remains an open question. For genetic analyses, genomic DNA extracted from a blood sample or a buccal swab from affected and unaffected members of families segregating hereditary hearing loss will be genetically screened with polymorphic markers (STRs or SNPs) for linkage to the known deafness loci. The hearing phenotype of children (>2 years old), adolescent and adult subjects will be assigned on the basis of performance from audiological examinations. Genomic DNA from families where deafness is found to be unlinked to the known deafness loci will then be used in genome wide screens with approximately 950,000 SNP markers distributed across the entire human genome to identify novel deafness loci. Alternatively, DNA samples from affected and unaffected individuals will undergo whole exome sequencing (WES) or whole genome sequencing (WGS) with a focus on potentially pathogenic variants located only in chromosomal regions of markers genetically linked to deafness. Subsequently, novel deafness genes will be positionally identified and their functions studied.

Outcome measures: Novel deafness loci and genes associated with hearing loss will be identified and will provide new insight into mechanisms required for sound transduction in humans. Data from this study is likely to be the basis of commercially available tests for early diagnosis and timely genetic counseling for at risk couples as well as the development of strategies to preserve hearing and prevent hearing loss.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Affected and unaffected members of families segregating deafness caused by genetic etiology.
* Adults must be able to provide informed consent.
* Adults must be able to provide informed consent for children who are at least two years of age
* All communities, ethnicities, and races as found in Pakistan.

EXCLUSION CRITERIA:

* Persons with non-genetic forms of hearing loss likely due to acquired causes such as an infection, head or noise trauma, or exposure to an ototoxic drug will not be included in this protocol
* Syndromic forms of inherited deafness are excluded if the gene for the disorder is known and there is no reason to believe the disorder is genetically heterogeneous.
* Subjects cannot provide informed consent or have a parent/guardian that cannot provide consent.
* Children under the age of two years will not be included in this study because an objective audiological examination such as an ABR analysis may require sedation, which is presently not feasible in Pakistan.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will ascertain subjects from consanguineous Pakistani families segregating hearing loss consisting of both nonsyndromic and syndromic forms of deafness of genetic etiology. Since a majority of Pakistani marriages are between first cousins, this tends to bring together the same recessive mutations for hearing loss with multiple affected individuals within single family lines, which is an advantage for this genetic study. A few years ago we stopped ascertaining families in India. We continue to ascertain both affected and unaffected Pakistani family members from age 2 years and up. Adults provide informed consent both for themselves and their children who agree to participate in this study. We will ascertain both genders and all Pakistani races and ethnicities.
Sampling Method: Probability Sample
Enrollment: 24000 (Estimated)
Dates: Start 2000-03-16 (Actual)

PRIMARY OUTCOMES:
To genetically map and identify additional genes causing hereditary hearing impairment in humans. | Ongoing
  -The number of novel deafness loci that we genetically map-The number of novel deafness genes we identify

SECONDARY OUTCOMES:
To study the function of genes in the auditory system | Ongoing
  -The structures and functions of the deafness genes revealed -Novel insight gained studying unrecognized hearing processes and pathophysiologies due to mutations of deafness genes we discover -Genotype/phenotype correlations that we identify that can be used to facilitate genetic diagnosis of hereditary hearing loss

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Friedman, Ph.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (1):
- University of Punjab, Lahore, Pakistan